CLINICAL TRIAL: NCT02660983
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Donepezil Hydrochloride (E2020) in Patients With Dementia Associated With Cerebrovascular Disease
Brief Title: A Study of Donepezil Hydrochloride in Patients With Dementia Associated With Cerebrovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-K082-418
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2018-05

CONDITIONS: Dementia Associated With Cerebrovascular Disease
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double Blind Phase: Placebo (Placebo Comparator): Participants will receive donepezil matching placebo, once daily in the evening during the double blind period.
  Interventions: Drug: Donepezil matching placebo
- Double Blind Phase: Donepezil (Experimental): Participants will receive donepezil 5 milligram (mg), once daily in the evening during the titration phase and then the dose will be increased to 10 mg at Week 4 during the double blind period. During the maintenance period, dose reduction to 5 mg/day will be permitted only when 10 mg/day is intolerable due to adverse events.
  Interventions: Drug: Donepezil hydrochloride
- Open-Label Extension Phase: Donepezil (Experimental): All participants who will complete the double-blind phase and want to continue the study participation, can be enrolled in the 24-week open-label extension phase. In this phase, treatment will be initiated at 5 mg/day, and the dose will be maintained until Week 6 (Day 28-42). After assessing clinical response during the period by examination, the dose can be increased to 10 mg/day. Dose reduction (from 10 mg/day to 5 mg/day) will be permitted when the investigator judges it difficult to continue the 10 mg/day administration. It will be possible to increase the dose to 10 mg/day again.
  Interventions: Drug: Donepezil hydrochloride

INTERVENTIONS:
Drug: Donepezil hydrochloride
  Other Names: E2020; Aricept
  Arms: Double Blind Phase: Donepezil
Drug: Donepezil matching placebo
  Arms: Double Blind Phase: Placebo
Drug: Donepezil hydrochloride
  Other Names: E2020; Aricept
  Arms: Open-Label Extension Phase: Donepezil

SUMMARY:
The primary objectives are to confirm that donepezil hydrochloride has superior efficacy compared with placebo in improving cognitive function, as measured by Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-cog), and to demonstrate that donepezil hydrochloride has superior efficacy compared with placebo in improving global function, as measured by Clinician's Interview-Based Impression of Change-plus Caregiver Input (CIBIC-plus), in patients with dementia associated with cerebrovascular disease (VaD).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel-group study with an open-label extension. The study consists of 3 phases; screening phase (1 to 4 weeks), double-blind phase (24 weeks), and Open-label extension phase (24 weeks). Participants, who have completed the double-blind phase and want to continue the study participation, can be enrolled in the 24-week open-label extension phase.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be eligible for inclusion in the study:

1. Male or female, age greater than or equal to (>=) 40 years at the time of informed consent.
2. Possible or probable dementia associated with cerebrovascular disease as defined by National Institute of Neurological Disorders and Stroke (NINDS) and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences (AIREN) criteria (NINDS-AIREN Criteria) with dementia of greater than 3 months duration.
3. Radiological evidence of cerebrovascular disease.
4. Mini-Mental Status Examination (MMSE) score is ≥ 10 and ≤ 24.
5. Clinical Dementia Rating (CDR) ≥ 1.
6. Outpatients who are physically healthy, and ambulatory or ambulatory-aided (i.e., walker, cane or wheelchair).
7. Written informed consent (IC) is obtained from the patient (if possible) and from the patient's legal guardian prior to being exposed to any study-related procedures. The caregiver must separately provide IC for his/her own participation in the study.
8. Patients having caregivers who submit written consent to cooperate with this study, have regular contact with the patient (i.e., an average of ≥ 4 hours/day and ≥ 3 days/week), provide patients' information necessary for this study, ensure the regular administration of assigned donepezil, as well as all concomitant therapies, at the correct dose, and escort the patients on required visits to study institution.
9. Comorbid medical conditions are clinically stable prior to Baseline, unless otherwise specified.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded:

1. Anti-dementia drug therapy (cholinesterase inhibitors or memantine) within 12 weeks prior to Screening.
2. Clinical and/or radiological evidence for other serious degenerative neurological disorders or neuropsychiatric disorders.
3. Known human immunodeficiency virus disease, neurosyphilis, or a history of significant head trauma followed by persistent neurological deficits or known structural brain abnormalities.
4. Hypothyroidism at Screening.
5. Vitamin B12 or folate deficiency at Screening.
6. Evidence of a new transient ischemic attack (TIA) or stroke that occurs within 12 weeks prior to Screening, even if the symptoms are minor and do not require hospitalization, are excluded.
7. Supine diastolic blood pressure ≥ 95 mmHg.
8. Complication of sick sinus syndrome, abnormal auricular and atrioventricular (AV) junction conductions (AV block, ≥ II ventricular block, etc.), or with a prolonged QT/QTc interval (> 450 ms) as demonstrated by a repeated electrocardiogram (ECG).
9. A history of life-threatening arrhythmias.
10. A history of malignant neoplasms treated within 5 years prior to study entry, current evidence of malignant neoplasm, recurrent, or metastatic disease.
11. A known or suspected history of drug or alcohol dependency or abuse.
12. Abnormal clinical laboratory values which are judged clinically significant by the investigator.
13. Patients who cannot swallow or who have difficulty swallowing whole tablets, as tablets should not be broken or crushed.
14. Known plan for elective surgery that would require general anesthesia and administration of neuromuscular blocking agents.
15. Pregnant women, lactating women, or women of child-bearing potential who don't agree to practice effective contraception throughout the entire study period and for 30 days after donepezil discontinuation, or who don't have a negative serum â-Human chorionic gonadotropin (HCG) test result or a negative urine pregnancy test result.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- South Korea (31):
  - Daegu, Buk-gu
  - Seongnam-si, Bundang-gu
  - Gwangju, Dong-gu
  - Seoul, Dongjak-gu
  - Seoul, Gangdong-gu
  - Seoul, Gangnam-gu
  - Chuncheon, Gangwon-do
  - Seoul, Gwangjin-gu
  - Anyang-si, Gyeonggi-do
  - Bucheon-si, Gyeonggi-do
  - Goyang-si, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Wonmi-gu, Gyeonggi-do
  - Changwon-si, Gyeongsangnam-do
  - Yangsan, Gyeongsangnam-do
  - Seoul, Jongro-gu
  - Daegu, Jung-gu
  - Incheon, Jung-gu
  - Seoul, Jungnang-Gu
  - Daegu, Nam-gu
  - Incheon, Namdong-gu
  - Busan, Seo-gu
  - Seoul, Seocho-gu
  - Seoul, Seodaemun-Gu
  - Seoul, Seongbuk-gu
  - Seoul, Seongdong-gu
  - Jongno-Gu, Seoul
  - Seoul, Songpa-Gu
  - Seoul, Yangcheon-gu
  - Seoul, Yeongdeungpo-gu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 32 investigative sites in Korea from 05 August 2013 to 21 December 2018.
Pre-assignment Details: A total of 425 participants were screened, of which 123 were screen failures and 302 were enrolled and randomized to receive study treatment. For Double Blind (DB) Phase both efficacy and safety data is presented while for Open Label Extension (OLE) Phase, only safety data is presented.
Groups:
- Placebo in DB Phase Then Donepezil in OLE Phase: Participants received placebo matched to donepezil 5 milligram (mg) tablet, orally, once daily in the evening for up to Week 4 in titration period, followed by placebo matched to donepezil 10 mg or 5 mg tablet, orally, once daily for up to Week 24 in maintenance period. Total duration of titration and maintenance period in Double Blind (DB) Phase was up to 24 weeks. Following completion of DB Phase, participant who had consent to continue their participation in the study entered the Open Label Extension (OLE) Phase and received donepezil 5 mg tablet, orally daily till Week 6 of OLE phase. After assessment of response, maximum dose permitted was 10 milligram per day (mg/day) up to Week 24 of OLE phase. Dose reduction to 5 mg/day was permitted upon investigator discretion.
- Donepezil in DB Phase Then Donepezil in OLE Phase: Participants received donepezil 5 mg, tablet, orally, once daily in the evening for up to Week 4 in titration period, followed by donepezil 10 mg, tablet, orally, once daily for up to Week 24 in maintenance period. Dose reduction to 5 mg/day was permitted only when 10 mg/day was intolerable due to an occurrence of adverse events of which the causal relationship with the donepezil was not ruled out. Total duration of titration and maintenance period in DB Phase was up to 24 weeks. Following completion of DB Phase, participant who had consent to continue their participation in the study entered the OLE Phase and received donepezil 5 mg tablet, orally daily till Week 6 of OLE phase. After assessment of response, maximum dose permitted was 10 mg/day up to Week 24 of OLE phase. Dose reduction to 5 mg/day was permitted upon investigator discretion.
Period: Double-blind (DB) Phase (24 Weeks)
Arm/Group | Placebo in DB Phase Then Donepezil in OLE Phase | Donepezil in DB Phase Then Donepezil in OLE Phase
Started | 154 | 148
Treated/Safety Set | 153 | 147
Completed | 130 | 122
Not Completed | 24 | 26
Not completed — Protocol Violation | 1 | 5
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Adverse Event | 8 | 9
Period: Open Label Extension Phase (24 Weeks)
Arm/Group | Placebo in DB Phase Then Donepezil in OLE Phase | Donepezil in DB Phase Then Donepezil in OLE Phase
Started | 86 (Eligible participants who consented to continue from DB phase to OLE phase.) | 75 (Eligible participants who consented to continue from DB phase to OLE phase.)
Safety Set | 86 | 75
Completed | 83 | 66
Not Completed | 3 | 9
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 1 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was the group of randomized participants who received at least one dose of study drug and had at least one postdose primary efficacy measurement.
Groups:
- Double Blind (DB) Phase: Placebo: Participants received placebo matched to donepezil 5 mg tablet, orally, once daily in the evening for up to Week 4 in titration period, followed by placebo matched to donepezil 10 mg or 5 mg tablet, orally, once daily for up to Week 24 in maintenance period. Total duration of titration and maintenance period in DB Phase was up to 24 weeks.
- Double Blind (DB) Phase: Donepezil: Participants received donepezil 5 mg, tablet, orally, once daily in the evening for up to Week 4 in titration period, followed by donepezil 10 mg, tablet, orally, once daily for up to Week 24 in maintenance period. Dose reduction to 5 mg/day was permitted only when 10 mg/day was intolerable due to an occurrence of adverse events of which the causal relationship with the donepezil was not ruled out. Total duration of titration and maintenance period in DB Phase was up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Double Blind (DB) Phase: Placebo | Double Blind (DB) Phase: Donepezil | Total
Number analyzed (Participants) | 146 | 137 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.96 (7.94) | 72.31 (7.06) | 72.64 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 48 | 103
  Male | 91 | 89 | 180
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 146 | 137 | 283

OUTCOME MEASURES:

1. Primary Outcome: Double Blind (DB) Phase: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) Score (LOCF) at Week 24
Description: The ADAS-Cog was a validated psychometric instrument that evaluates memory (word recall, word recognition), attention, reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). The ADAS-cog scores range from 0 to 70, with negative change from baseline indicating clinical improvement. LOCF=last observation carried forward.
Time Frame: Baseline and Week 24
Population: The FAS, LOCF, included all randomized participants who received at least one dose of study drug and had at least one postdose primary efficacy measurement. Overall number of participants analyzed included participants who were evaluable at a particular time point for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double Blind (DB) Phase: Placebo | Double Blind (DB) Phase: Donepezil
Number analyzed (Participants) | 144 | 133
score on a scale | -2.06 (0.42) | -2.64 (0.44)
Statistical Analysis 1: Comparison: Double Blind (DB) Phase: Placebo vs Double Blind (DB) Phase: Donepezil; Test type: Superiority; p = 0.3455, ANCOVA; Difference in least square (LS) means = -0.58, 95% CI 2-sided [-1.79 to 0.63]

2. Primary Outcome: Double Blind (DB) Phase: Clinicians Interview-based Impression of Change-plus Caregiver Input (CIBIC-plus) Score (LOCF)
Description: The CIBIC-plus rates change in global functioning relative to baseline on a scale. The score ranges from 1 (Marked improvement) to 7 (Marked worsening). A score of "4" represents no change from baseline. LOCF=last observation carried forward.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double Blind (DB) Phase: Placebo | Double Blind (DB) Phase: Donepezil
Number analyzed (Participants) | 146 | 135
score on a scale | 3.85 (0.07) | 3.73 (0.07)
Statistical Analysis 1: Comparison: Double Blind (DB) Phase: Placebo vs Double Blind (DB) Phase: Donepezil; Test type: Superiority; p = 0.2570, ANCOVA; Difference in LS means = -0.12, 95% CI 2-sided [-0.32 to 0.09] — LS mean of Donepezil group - LS mean of Placebo (when the difference of LS mean scores were less than 0, considered as demonstrated hypothesis), analyzed with ANCOVA model with baseline (CIBIS) as covariate and treatment as main effect

3. Secondary Outcome: Double Blind (DB) Phase: Change From Baseline in Mini-mental State Examination (MMSE) Score (LOCF) at Week 24
Description: MMSE is a well-known, gold standard test for measuring the cognitive state of dementia participants. It includes items evaluating orientation to time and place, recall of objects, attention, language, and conversational abilities. The total score ranges from 0 (most impaired) to 30 (no impairment). The lower score means severe cognitive deficit. A positive change score indicated improvement from baseline. LOCF=last observation carried forward.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double Blind (DB) Phase: Placebo | Double Blind (DB) Phase: Donepezil
Number analyzed (Participants) | 146 | 136
score on a scale | 0.59 (0.22) | 1.23 (0.22)
Statistical Analysis 1: Comparison: Double Blind (DB) Phase: Placebo vs Double Blind (DB) Phase: Donepezil; Test type: Superiority; p = 0.0396, ANCOVA; Difference in LS means = 0.65, 95% CI 2-sided [0.03 to 1.26]

4. Secondary Outcome: Double Blind (DB) Phase: Change From Baseline in Executive Function Test (Korean Trail Making Test Elderly [K-TMT-e]) Score (LOCF) at Week 24
Description: The trail making test (TMT) was an evaluation tool used to assess the cognitive function, especially for executive function. The K-TMT-e has two parts that are referred to as part A (component: serial numbers) and part B (component: serial numbers and days). The K-TMT-e was a timed test and the goal was to complete the tests accurately and as quickly as possible. Higher scores reveal greater impairment. K-TMT-e Score was measured as time taken by participants to complete goal. LOCF=last observation carried forward.
Time Frame: Baseline and Week 24
Population: The FAS, LOCF, included all randomized participants who received at least one dose of study drug and had at least one postdose primary efficacy measurement. Number analyzed signifies participants who were evaluable at a particular part of study for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Double Blind (DB) Phase: Placebo | Double Blind (DB) Phase: Donepezil
Number analyzed (Participants) | 146 | 137
seconds
  Part A: number analyzed (Participants) | 134 | 126
  Part A | -5.10 (4.38) | -12.82 (4.52)
  Part B: number analyzed (Participants) | 127 | 122
  Part B | 1.16 (5.41) | -13.73 (5.52)
Statistical Analysis 1: Comparison: Double Blind (DB) Phase: Placebo vs Double Blind (DB) Phase: Donepezil; Part A; Test type: Superiority; p = 0.2213, ANCOVA; Difference in LS means = -7.73, 95% CI 2-sided [-20.13 to 4.68]
Statistical Analysis 2: Comparison: Double Blind (DB) Phase: Placebo vs Double Blind (DB) Phase: Donepezil; Part B; Test type: Superiority; p = 0.0551, ANCOVA; Difference in LS means = -14.88, 95% CI 2-sided [-30.10 to 0.33]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 30 days after the last dose of study drug (up to 52 weeks [DB Phase: From the first dose of study drug till Week 24; OLE Phase: Post Week 24 till Week 52])
Description: Safety analysis set: all participants who signed informed consent received at least 1 dose of study drug and had at least 1 post-dose safety assessment. If adverse event was non-serious adverse event in DB Phase but became serious adverse event during OLE Phase, the adverse event was also analyzed as serious adverse event in OLE Phase.
Groups:
- Open Label Extension (OLE) Phase: Donepezil: Participants who completed DB phase and consented to continue their participation in the study, were enrolled in OLE phase. In OLE phase, initially all participants received donepezil 5 mg tablet, orally daily till Week 6 of OLE phase. After assessment of response, maximum dose permitted was 10 mg/day up to Week 24 of OLE phase. Dose reduction to 5 mg/day was permitted upon investigator discretion.
Arm/Group | Double Blind (DB) Phase: Placebo | Double Blind (DB) Phase: Donepezil | Open Label Extension (OLE) Phase: Donepezil
All-Cause Mortality (participants affected / at risk) | 1/153 | 1/147 | 2/161
Serious Adverse Events (participants affected / at risk) | 24/153 | 18/147 | 12/161
Other Adverse Events (participants affected / at risk) | 73/153 | 86/147 | 63/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB) Phase: Placebo (N=153) | Double Blind (DB) Phase: Donepezil (N=147) | Open Label Extension (OLE) Phase: Donepezil (N=161)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion 1 (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Infarction (Vascular disorders) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB) Phase: Placebo (N=153) | Double Blind (DB) Phase: Donepezil (N=147) | Open Label Extension (OLE) Phase: Donepezil (N=161)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 10 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 1
Vomiting (Gastrointestinal disorders) | 1 | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 2
Pyrexia (General disorders) | 1 | 1 | 0
Oedema (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 6 | 4
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Periodontitis (Infections and infestations) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 2
Blood pressure increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 11 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 9 | 5
Dizziness (Nervous system disorders) | 6 | 5 | 3
Paraesthesia (Nervous system disorders) | 1 | 1 | 2
Poor quality sleep (Nervous system disorders) | 1 | 1 | 1
Tremor (Nervous system disorders) | 1 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 7 | 1
Conduct disorder (Psychiatric disorders) | 0 | 2 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 2
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0
Incontinence (Renal and urinary disorders) | 1 | 1 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Bladder dysfunction (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Tenderness (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Trichiasis (Eye disorders) | 0 | 0 | 1
Astigmatism (Eye disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT02660983/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02660983/SAP_001.pdf